CLINICAL TRIAL: NCT05865119
Title: OPTImal Treatment of Sinus VENOSUS Defect - Efficacy and Safety of Transcatheter Correction Compared to Surgical Treatment in Patients With Sinus Venosus Defect
Brief Title: OPTImal Treatment of Sinus VENOSUS Defect
Acronym: OPTIVENOSUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A01507-36
Record Dates: First submitted 2023-03-14; First posted 2023-05-18 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Sinus Venosus Defect; Congenital Heart Disease; Sinus Venosus Atrial Septum Defect
Keywords: congenital heart disease; sinus venosus; stent; surgery; comparative study; 3D printing; simulation; rare disease; optimus; catheterization
MeSH Terms: conditions — Atrial Septal Defect Sinus Venosus; Heart Defects, Congenital; Rare Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endovascular (Experimental): Transcatheter correction of a SVD with an OPTIMUS covered stent
  Interventions: Device: OPTIMUS covered stent
- surgery (Active Comparator): Surgical correction of a SVD
  Interventions: Procedure: Surgical correction of a SVD

INTERVENTIONS:
Device: OPTIMUS covered stent — The procedure involves placement of a long and large balloon-expandable covered stent in the superior vena cava that tunnels the abnormal pulmonary venous return to the left atrium.
  Arms: endovascular
Procedure: Surgical correction of a SVD — Under cardiopulmonary bypass and open heart surgery, surgical correction of SVD either using single patch, double patch or Warden techniques
  Arms: surgery

SUMMARY:
Sinus venosus defect (SVD) accounts for 10% of atrial septal defects and is characterized by an anomalous pulmonary venous return in the superior vena cava associated with a high situated atrial septal defect. Since 2013, transcatheter correction of this congenital heart disease has emerged as a new treatment option. The procedure involves placement of a covered stent in the superior vena cava that tunnels the anomalous pulmonary venous return to the left atrium. Preliminary results are limited but promising.

The devices to be used depend on anatomic considerations. XXL stents than 70mm are often required. Today, the availability of CE marked stents is limited. There have been recent reports of successful corrections with the specifically developed Optimus XXL 100mm covered stent (ANDRATEC) with compassionate approval from the Agence Nationale de Sûreté du Médicament in France. Setting up a feasibility study to investigate the use of medical devices in this indication was required.

The objective of this project is to study the feasibility, efficacy and safety of the Optimus stent in this newly developed transcatheter procedure, in comparison with the gold-standard surgical method. A French national multicenter comparative cohort study including all eligible patients referred for transcatheter correction of SVD was designed. The feasibility of the transcatheter procedures will be investigated beforehand by virtual digital simulation and simulation on a 3D printed model. The procedures will then be performed in centers of the M3C network for complex congenital heart diseases (CARDIOGEN). The primary endpoint will be a composite of efficacy, defined as complete occlusion of the shunt, and safety, defined as the absence of major events at 6 months. The secondary endpoints will be anatomical, functional and psychosocial (quality of life).

It is expected that transcatheter treatment gives comparable results to surgery on the primary endpoint. This could justify the further development of this procedure as an alternative to surgery and facilitate the validation of dedicated equipment.

DETAILED DESCRIPTION:
OPTIVENOSUS will be offered to patients who have an correction of SVD. A pre-therapeutic assessment will be prescribed with a CT scan and MRI, followed by a complementary assessment with a 6-minute walk test, a functional cardiorespiratory examination, a Holter and an ECG.

In addition, the images from the CT scan carried out during the pre-therapeutic assessment will be transferred to a secure platform approved for hosting health data. These images will be the subject of a 3D reconstruction.

Then a multidisciplinary consultation meeting held by paediatric cardiologists, specialists in adult congenital heart disease, surgeons and interventional cardiologists will be held to assess whether or not the patient is ineligible for surgery and whether or not the patient is eligible for transcatheter correction of SVD on the basis of the imaging examinations and the clinical assessment.

During this meeting, the imaging core lab and the experts will give their opinion on the feasibility of the endovascular procedure.

The criteria considered for ineligibility for surgery will include

* Comorbidities
* Complications (rhythm disorders, heart failure, pulmonary hypertension).
* Age of the patient
* Anatomical considerations

The criteria considered for eligibility for percutaneous treatment are:

* Ineligibility for surgery
* An adult patient with a compatible anatomy (distance between the upper edge of the anomalous pulmonary venous return and the lower edge of the innominate venous trunk > 2cm allowing sufficient stent attachment in the SVD; a diameter of the atrial septal defect >10mm allowing redirection of flow from the anomalous pulmonary venous return to the left atrium without restriction and a position of the anomalous pulmonary veins allowing redirection of flow to the left atrium without obstruction by the stent in digital simulation). These 3 elements will be analysed on the injected scanner and then confirmed by the scanner simulation, the 3D printed model and the simulation of the procedure on an experimental test bench.

If the patient is eligible for the endovascular approach, a bench simulation of the endovascular procedure will be performed.

A simulation of the endovascular procedure is performed on a test bench in the hybrid room of the Marie Lannelongue Hospital. The test bench consists of a 3D model of the heart that corresponds exactly to the patient's anatomy, produced using CT images.

The simulation allows on the one hand to confirm the feasibility of transcatheter correction of SVD and on the other hand to define the characteristics in terms of diameter and length of the necessary devices (stent and balloons) for the procedure in order to have a personalized approach.

The simulation session will take place in the presence of the referring interventional cardiologists.

All patients, regardless of the mode of correction of SVD, will have the same follow-up at D7, 1 month, 6 months and then every year for 5 years with an echographic control and a clinical evaluation

ELIGIBILITY:
Inclusion Criteria:

* from 12 years of age
* SVD with right ventricular end-diastolic volume dilatation (RV EDV) on imaging (echocardiography and/or MRI), defined by the guidelines as RV EDV greater than 112mL/m2 for women and 121 mL/m2 for men.
* With an indication for atrial septal defect correction, indicated at a medical-surgical meeting according to the ESC 2020 guideline criteria
* Adult patients who received informed information about the study and signed a consent to participate in the study
* Minor patients, no opposition from both holders of parental authority to data processing.
* Patient agreeing to be followed for the duration of the study
* Affiliated or beneficiary of a social security plan NB: Minor patients will only be considered eligible for the surgical procedure and will be studied descriptively.

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under judicial protection
* Pregnant or breastfeeding woman
* Patient already included in an interventional research protocol

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-05-12 (Estimated); Study Completion 2029-05-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants meeting the primary net criteria in the 2 groups | At six month
  Number of participants (%) with complete occlusion of the shunt AND absence of a major procedure-related event (death or open-heart surgery).

SECONDARY OUTCOMES:
Number of participants meeting the Safety and technical success criteria at 1 month | At one month
  - Number of participants (%) with Technical success rate of the correction procedure defined by correction of Abnormal Pulmonary Venous Return and shunt occlusion AND absence of each of the following complications: ECMO, dialysis, stroke, rhythm disorder requiring drug or electrical intervention, severe conduction disorder requiring pace maker AND absence of re-hospitalization or prolongation of initial hospitalization due to a procedure-related Serious Adverse Event
Difference in functional capacity before versus after intervention | At six months
  Change in baseline and 6-month 6 minutes walking test (in meters)
Difference in NYHA status before versus after intervention | At six months
  Change in baseline and 6-month NYHA score (score from 0 to 4 O the best status 4 the worst functional class)
Number of participants meeting the safety criteria at one year | At one year
  Number of participants (%) with percutaneous or surgical re-intervention, or stroke or conduction rhythm disorder requiring pacemaker placement.
Number of participants meeting the safety criteria at 2 years | At two years
  Number of participants (%) with percutaneous or surgical re-intervention, or stroke or conduction rhythm disorder requiring pacemaker placement.
Number of participants meeting the safety criteria at three years | At three years
  Number of participants (%) with major complications related to the heart disease
Number of participants meeting the safety criteria at four years | At four years
  Number of participants (%) with major complications related to the heart disease
Number of participants meeting the safety criteria at five years | At five years
  Number of participants (%) with major complications related to the heart disease

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien HASCOËT, Principal Investigator — Hôpital Marie Lannelongue; Alban-Elouen BARUTEAU, Principal Investigator — Nantes University Hospital
Locations (13):
- France (13):
  - CHU Bordeaux, Bordeaux
  - Hospices Civils de Lyon, Bron
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - Sébastien HASCOËT, Le Plessis-Robinson
  - CHU Lille, Lille
  - Hôpitaux universitaire de Marseille, Marseille
  - CHU Nantes, Nantes
  - CHU Necker APHP Paris, Paris
  - HEGP Paris, Paris
  - CHU Toulouse, Toulouse
  - Clinique Pasteur, Toulouse, Toulouse
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Batteux C, Azarine A, Karsenty C, Petit J, Ciobotaru V, Brenot P, Hascoet S. Sinus Venosus ASDs: Imaging and Percutaneous Closure. Curr Cardiol Rep. 2021 Aug 19;23(10):138. doi: 10.1007/s11886-021-01571-7. PMID 34410510
- [Background] Batteux C, Ciobotaru V, Bouvaist H, Kempny A, Fraisse A, Hascoet S. Multicenter experience of transcatheter correction of superior sinus venosus defect using the covered Optimus XXL stent. Rev Esp Cardiol (Engl Ed). 2023 Mar;76(3):199-201. doi: 10.1016/j.rec.2022.08.004. Epub 2022 Aug 30. No abstract available. English, Spanish. PMID 36055641
- [Background] Rosenthal E, Qureshi SA, Jones M, Butera G, Sivakumar K, Boudjemline Y, Hijazi ZM, Almaskary S, Ponder RD, Salem MM, Walsh K, Kenny D, Hascoet S, Berman DP, Thomson J, Vettukattil JJ, Zahn EM. Correction of sinus venosus atrial septal defects with the 10 zig covered Cheatham-platinum stent - An international registry. Catheter Cardiovasc Interv. 2021 Jul 1;98(1):128-136. doi: 10.1002/ccd.29750. Epub 2021 May 7. PMID 33909945
- [Background] Batteux C, Meliani A, Brenot P, Hascoet S. Multimodality fusion imaging to guide percutaneous sinus venosus atrial septal defect closure. Eur Heart J. 2020 Dec 7;41(46):4444-4445. doi: 10.1093/eurheartj/ehaa292. No abstract available. PMID 32428931
- [Background] Haddad RN, Bonnet D, Gewillig M, Malekzadeh-Milani S. Modified safety techniques for transcatheter repair of superior sinus venosus defects with partial anomalous pulmonary venous drainage using a 100-mm Optimus-CVS(R) covered XXL stent. Catheter Cardiovasc Interv. 2022 Apr;99(5):1558-1562. doi: 10.1002/ccd.30136. Epub 2022 Feb 22. PMID 35192742
- [Background] Baruteau AE, Jones MI, Butera G, Qureshi SA, Rosenthal E. Transcatheter correction of sinus venosus atrial septal defect with partial anomalous pulmonary venous drainage: The procedure of choice in selected patients? Arch Cardiovasc Dis. 2020 Feb;113(2):92-95. doi: 10.1016/j.acvd.2019.09.014. Epub 2020 Feb 11. No abstract available. PMID 32057661
- [Derived] Batteux C, Ciobotaru V, Haddad RN, Houeijeh A, Karsenty C, Bouzguenda I, Roussin R, Combes N, Bakloul M, Aldebert P, Dion F, Lefort B, Bosser G, Bonnet D, Fraisse A, Bouvaist H, Hoerer J, Moceri P, Godart F, Lenoir M, Dauphin C, Radojevic J, Thambo JB, Lecerf F, Hache O, Chevalier D, Beaussier H, Aubrege L, Azarine A, Decante B, Chatellier G, Ladouceur M, Baruteau AE, Henaine R, Albenque G, Hascoet S. Safety and efficacy of transcatheter correction of sinus venosus defect using 70-100mm-long partially covered Optimus-CVS(R) XXL stents compared with surgery: The OPTIVENOSUS study design. Arch Cardiovasc Dis. 2025 Sep;118(8-9):497-507. doi: 10.1016/j.acvd.2025.05.003. Epub 2025 May 29. PMID 40571458
- See also: Baruteau AE, Jones MI, Butera G, Qureshi SA, Rosenthal E. Transcatheter correction of sinus venosus atrial septal defect with partial anomalous pulmonary venous drainage: The procedure of choice in selected patients? Arch Cardiovasc Dis. 2020 — https://pubmed.ncbi.nlm.nih.gov/32057661/
- See also: Batteux C, Azarine A, Karsenty C, Petit J, Ciobotaru V, Brenot P, Hascoet S. Sinus Venosus ASDs: Imaging and Percutaneous Closure. Curr Cardiol Rep. 2021 Aug 19;23(10):138. doi: 10.1007/s11886-021-01571-7 — https://pubmed.ncbi.nlm.nih.gov/34410510/
- See also: Batteux C, Ciobotaru V, Bouvaist H, Kempny A, Fraisse A, Hascoet S. Multicenter experience of transcatheter correction of superior sinus venosus defect using the covered Optimus XXL stent. Rev Esp Cardiol (Engl Ed). 2023 Mar;76(3):199-201. — https://pubmed.ncbi.nlm.nih.gov/36055641/
- See also: Rosenthal E, Qureshi SA, Jones M, Butera G, Sivakumar K, Boudjemline Y, Hijazi ZM, Almaskary S, Ponder RD, Salem MM, Walsh K, Kenny D, Hascoet S, Berman DP, Thomson J, Vettukattil JJ, Zahn EM. Correction of sinus venosus atrial septal defects with the 10 — https://pubmed.ncbi.nlm.nih.gov/33909945/
- See also: Batteux C, Meliani A, Brenot P, Hascoet S. Multimodality fusion imaging to guide percutaneous sinus venosus atrial septal defect closure. Eur Heart J. 2020 Dec 7;41(46):4444-4445. doi: 10.1093/eurheartj/ehaa292. No abstract available. — https://pubmed.ncbi.nlm.nih.gov/32428931/
- See also: Haddad RN, Bonnet D, Gewillig M, Malekzadeh-Milani S. Modified safety techniques for transcatheter repair of superior sinus venosus defects with partial anomalous pulmonary venous drainage using a 100-mm Optimus-CVS(R) covered XXL stent. — https://pubmed.ncbi.nlm.nih.gov/35192742/